CLINICAL TRIAL: NCT01218399
Title: A Randomized, Blinded, Single-center Study in Mild to Moderate Asthmatics Over the Age of 12 Years Who Have a Viral-mediated Exacerbation and Are Treated With Symbicort or Pulmicort Flexhaler
Brief Title: Use of Symbicort or Pulmicort to Treat Viral-mediated Asthma Exacerbations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Kari Christine Nadeau, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU-10042010-7010; IRB 15128
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Active Comparator): Combination of budesonide and formoterol. Medications are given according to the package insert and manufacturer's instructions.
  Participants that develop a viral upper respiratory illness which induces an asthma exacerbation.within the specified period following enrollment, are randomly assigned 1:1 to either study arm. 5 participants were randomly assigned to the Symbicort study arm.
  Interventions: Drug: Symbicort
- Placebo Comparator: Budesonide (Placebo Comparator): Control of budesonide alone. Medication was given according to the package insert and manufacturer's instructions.
  Participants that develop a viral upper respiratory illness which induces an asthma exacerbation.within the specified period following enrollment, are randomly assigned 1:1 to either study arm. 5 participants were randomly assigned to the Budesonide study arm.
  Interventions: Drug: Symbicort

INTERVENTIONS:
Drug: Symbicort
  Other Names: Budesonide

SUMMARY:
This is an investigator-initiated study in which Dr. Nadeau wrote the protocol and received funding from an Astra Zeneca grant to direct, perform, and monitor the study on her own with Stanford staff. We hypothesize that the budesonide/formoterol combination improves the efficacy of budesonide alone.

DETAILED DESCRIPTION:
The study was designed such that 30 participants would be consented/enrolled into the trial. The intervention would only be applied if the participant developed a viral illness that met eligibility criteria during the study period.

Only 10 of the 30 ppt. consented/enrolled developed a virus and were then treated according to study arm.

A more detailed description can be obtained by contacting Astra Zeneca

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered for inclusion in this study based on meeting all of the following criteria:

1. Male or female, aged 12 to 65 years
2. Subjects with mild to moderate asthma as determined by NHLBI 2007 guidelines
3. Subjects with exacerbation of their asthma symptoms by NHLBI 2007 guidelines
4. IgE level at study entry less than 50 IU/mL
5. Men and women of reproductive potential who document use of adequate contraception during the study and for 3 months after the conclusion of treatment with study drug/placebo
6. Historical documentation of asthma in the patient's medical record. The patient should have 6 months or more of asthma medication and management by a Stanford physician.
7. Women of childbearing potential who have a negative pregnancy test (urine or serum) at the time of study entry
8. Subject's guardians who are capable of understanding the purpose and risks of the study and who sign a statement of informed consent for the study

Exclusion Criteria:

Subjects will be ineligible for this study based on any one of the following criteria:

1. With a chronic or acute disease that might interfere with the evaluation of Symbicort or Pulmicort Flexhaler therapy
2. Pregnancy or lactation
3. Current or prior malignancies (excluding non-melanoma skin carcinoma or carcinoma in situ of the cervix that has been adequately treated)
4. History of infection with human immunodeficiency virus (HSC-1), hepatitis B virus (HBV), or hepatitis C virus (HCV); or Hepatitis A virus (HAV)
5. Infections that require intravenous antibiotic therapy
6. Significant organ dysfunction, including cardiac, renal, liver, CNS, pulmonary, vascular, gastrointestinal, endocrine, or metabolic (e.g., creatinine >1.6 mg/dL; ALT or AST > 1.5x the upper limit of normal; history of myocardial infarction, congestive heart failure, or arrhythmias within 6 months prior to study entry)
7. Treatment with a humanized or chimeric antibody therapy within 4 weeks prior to study entry
8. Treatment with any investigational drugs or therapies within 2 weeks prior to study entry
9. Any use of oral, systemic corticosteroids within 2 weeks prior to study entry

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Christine Nadeau, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants that contract a viral upper respiratory illness which induces an asthma exacerbation and meets eligibility criteria will be randomized at Day 1 to either Symbicort or Budesonide in a 1:1 randomization. 5 participants were randomly assigned to the Symbicort study arm, and 5 participants were assigned to the Budesonide study arm.
Groups:
- Symbicort: Combination of budesonide and formoterol
  Symbicort will be given as per product insert (2 puffs twice daily of 160/4.5 Budesonide/formoterol)
- Budesonide: Control of budesonide alone
  Pulmicort Flexhaler will be given as per product insert (2 puffs twice daily of 160 mcg)
Period: Overall Study
Arm/Group | Symbicort | Budesonide
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Symbicort: combination of budesonide and formoterol
  Symbicort vs Budesonide in treating acute respiratory illness: use of either symbicort or budesonide
- Budesonide: control of budesonide alone
  Symbicort vs Budesonide in treating acute respiratory illness: use of either symbicort or budesonide
- Total: Total of all reporting groups
Arm/Group | Symbicort | Budesonide | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (5) | 25 (6) | 24 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Forced Expiratory Volume in One Second (FEV1)
Description: Asthma symptoms scores reported as measure of FEV1 - Forced Expiratory Volume in one second
  * FEV1 is given which is a standard outcome in asthma studies and is validated by the NIH (NHLBI)
  * FEV1 of less than 80 is indicative of severe asthma, 80-90 is moderate asthma, over 90 is mild asthma
  http://www.med.umich.edu/1info/FHP/practiceguides/asthma/EPR-3_pocket_guide.pdf
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: % FEV1
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5 | 5
% FEV1 | 90 (13) | 88 (14)

2. Secondary Outcome: Adverse Events
Description: Number of adverse events as per MEDRA terms
Time Frame: 1 week
Measure: Number; unit: Number adverse events
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5 | 5
Number adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Data was collected for a year
Arm/Group | Symbicort | Budesonide
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact the sponsor Astra Zeneca for the agreement